CLINICAL TRIAL: NCT00530517
Title: A Multi-Center, Open-Label, Single-dose, Single-Arm Study to Evaluate the Usability of Subcutaneously Administered Sumatriptan Delivered Via the Intraject® System in Adult Patients During Acute Migraine Attack
Brief Title: A Study on the Usability of the Needle-free Intraject® System in Adult Patients During Acute Migraine Attack
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Stephen J. Farr, Ph.D/ President and COO, Zogenix, Inc
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZX001-0701
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2008-02

CONDITIONS: Migraine Headache
Keywords: migraine; sumatripatan
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Intraject Sumatriptan

INTERVENTIONS:
Device: Intraject Sumatriptan — needle-free, single use, disposable, subcutaneous delivery system pre-filled with 6mg Sumatriptan

SUMMARY:
Intraject is a needle-free, single use, disposable, subcutaneous delivery system pre-filled with 6mg Sumatriptan to be used by patients to treat acute migraine treatment. Study participation will last one month and include 2 doctor visits and 2-4 phone calls.

DETAILED DESCRIPTION:
This study will evaluate how patients will interact with the needle-free Intraject system during actual self-administration to the abdomen or thigh for treatment of migraine headache while outside the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine with an average of ≥2 to ≤6 attacks/month
* Female subjects of child-bearing potential must agree to use acceptable birth control
* Have abdominal or thigh injection sites that have sufficient subcutaneous tissue for needle-free injection
* Fluent in the spoken and written English language
* Provide written informed consent to participate in the study and be willing to comply with the study procedures
* Access to a telephone for call center interactions

Exclusion Criteria:

* A history, symptoms, or signs of ischemic cardiac, cerebrovascular, or peripheral vascular syndromes including ischemic or vasospastic coronary artery disease
* Other significant underlying cardiovascular diseases including uncontrolled hypertension
* Hemiplegic or basilar migraine
* A history or diagnosis of severe hepatic or renal impairment
* A history of epilepsy or seizure or other serious neurologic condition
* A history of allergy, anaphylaxis, or hypersensitivity to sumatriptan or any of its components or similar drugs
* A history of scleroderma (systemic sclerosis) or any skin condition that may adversely affect the injection or absorption of subcutaneously administered medications
* Tattoos in the thigh or abdominal area that are large enough to restrict injection site selection and/or evaluation
* Birthmark or other significant skin discoloration in the thigh or abdominal area large enough to restrict injection site selection and/or evaluation
* Pregnancy or breast-feeding
* Have participated in a clinical trial or receipt of an experimental therapy within 30 days prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the usability of sumatriptan delivered subcutaneously via the Intraject system in adult patients during acute migraine attack | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brandes, MD, Principal Investigator — Nashville Neuroscience Group
Locations (4):
- United States (4):
  - Chicago, Illinois
  - Springfield, Missouri
  - St Louis, Missouri
  - Nashville, Tennessee